CLINICAL TRIAL: NCT05281965
Title: A Clinical Study Evaluating the Efficacy and Safety of Retinoic Acid in Patients With 15q11-q13 Duplication Syndrome
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-0438
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Autism; Treatment Adherence; Retinoic Acid; Dup15Q Syndrome
MeSH Terms: conditions — Autistic Disorder; Treatment Adherence and Compliance | interventions — Tretinoin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Drug: Retinoic acid
- Placebo group (Placebo Comparator)
  Interventions: Drug: Retinoic acid

INTERVENTIONS:
Drug: Retinoic acid — Retinoic acid oral

SUMMARY:
Autism Spectrum Disorders (ASD), with its core symptoms of communication and repetitive behaviors, is a serious neurodevelopmental disorder common in childhood and affects about 1% of children. So far, autism remains a clinical dilemma with no effective therapy.

The most common chromsomal ability among ASD patients is 15q11-13q duplication syndrome(dup15q syndrome).Clinical phenotypes of dup15q syndrome include autism, mental retardation, epilepsy (usually refractory epilepsy, often manifested as infantile spasm), congenital heart disease, mild facial abnormalities, etc.

UBE3A is one of the most important genes in the 15q11-q13 region.Biochemistry and molecular biology of the Chinese Academy of Sciences Hu Ronggui group found a new kind of autism in mechanisms and potential therapeutic targets - describe the ubiquitin ligase UBE3A protein and retinoic acid.Previous studies have shown that the basis of the relevant treatment measures can effectively relieve the mouse model of autism characteristics. Therefore, retinoic acid supplementation in the treatment of dup15q syndrome is a potential therapeutic target.

ELIGIBILITY:
Inclusion Criteria:

1. Between 6 and 18 years old
2. Clinical diagnosis + scale diagnosis of autism (1) Clinical diagnosis: clinical diagnosis was made by 2 experienced doctors according to the medical history provided by the caregivers and the diagnostic criteria of ASD in DSM-V; (2) Scale diagnosis: The diagnostic assessment was conducted by highly qualified practitioners taking the ADOS-2 score, Restricted Behabior (RRB) and Social Affect (SA) scores. The scores were converted to standardized severity scores (CSS) for three diagnoses of non-spectrum disorders, autism and autism spectrum disorders.
3. Genetics: 15q11-13 duplicates diagnosed by SNP-Array or A-CGH microarray, including UBE3A gene

Exclusion Criteria:

1. A history of acute or chronic infection within the last 3 months
2. There are still active seizures within the past 1 year
3. Have taken vitamin and/or mineral supplements within the last 6 months
4. A history of chronic diseases, including abnormal liver function, abnormal kidney function, and abnormal thyroid function;

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
ADORS-2 | 3 months，6 months，9 months，12 months
  The primary outcome measure was changes in the social core symptom of ASD assessed using the social reciprocity score of Autism Diagnostic Observation Schedule (ADOS)39 module 4 (range: 0-14, higher values represent worse outcomes) between the baseline and end point of each administration period.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Zhejiang University, Hangzhou, Zhejiang
  - Miao pu, Hangzhou

IPD SHARING:
Plan to Share IPD: Undecided